CLINICAL TRIAL: NCT02708862
Title: Comparison of Emergency Department Preoxygenation Techniques in Healthy Volunteers
Brief Title: Four Methods of Pre-oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Preox
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoxygenation (Experimental): All participants were enrolled in a single arm in which they underwent 4 interventions in series: 1) Simple mask at 60 L/min for 3 minutes 2) Non-rebreather at 15 L/min for 3 min 3) Non-rebreather at 60 L/min for 3 minutes 4) Bag valve mask at 15 L/min for 3 minutes
  Interventions: Device: Preoxygenation

INTERVENTIONS:
Device: Preoxygenation — After 3 minutes of oxygen supplementation (preoxygenation), with each of the devices listed below, the exhaled oxygen content will be measured. All participants were enrolled in a single arm in which they underwent 4 interventions in series: 1) Simple mask at 60 L/min for 3 minutes 2) Non-rebreather at 60 L/min for 3 min 3) Non-rebreather at 15 L/min for 3 minutes 4) Bag valve mask at 15 L/min for 3 minutes

SUMMARY:
Four methods of preoxygenation will be compared in healthy volunteers

DETAILED DESCRIPTION:
After informed consent, each volunteer will undergo the following techniques:

Simple mask at "flush" flow (40-60 L/min) Non-rebreather mask at 15 L/min Non-rebreather mask at 60 L/min Bag valve mask with one way exhalation valve at 15 L/min

After 3 minutes, the exhaled oxygen will be measured with an oxygen sensor

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old

Exclusion Criteria:

* Any active respiratory pathology (asthma, chronic obstructive pulmonary disease, other lung disease, smoking history more than 5 years)
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Driver BE, Prekker ME, Kornas RL, Cales EK, Reardon RF. Flush Rate Oxygen for Emergency Airway Preoxygenation. Ann Emerg Med. 2017 Jan;69(1):1-6. doi: 10.1016/j.annemergmed.2016.06.018. Epub 2016 Aug 10. PMID 27522310

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 26 total subjects; each did all 4 arms.
Groups:
- Preoxygenation: All participants were enrolled in a single arm in which they underwent 4 interventions in series: 1) Simple mask at 60 L/min for 3 minutes 2) Non-rebreather at 60 L/min for 3 min 3) Non-rebreather at 60 L/min for 3 minutes 4) Bag valve mask at 15 L/min for 3 minutes
Period: Overall Study
Arm/Group | Preoxygenation
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preoxygenation
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Oxygen Concentration
Description: Subjects will blow into an oxygen sensor after each method (arm). The primary outcome will be a non-inferiority test between bag valve mask and non-rebreather at 60 L/min. The remaining tests will be completed for comparison, but not part of formal statistical testing.
Time Frame: Immediately after 3 minutes of oxygen supplementation
Measure: Mean (95% Confidence Interval); unit: % FeO2
Arm/Group | Preoxygenation
Number analyzed (Participants) | 26
% FeO2
  Simple mask at 60 L/min for 3 minutes | 72 [69 to 76]
  Non-rebreather at 60 L/min for 3 min | 86 [84 to 88]
  Non-rebreather at 15 L/min for 3 min | 54 [50 to 57]
  Bag valve mask at 15 L/min for 3 minutes | 77 [74 to 81]

ADVERSE EVENTS:
Groups:
- Simple Mask: Simple mask at 60 L/min for 3 minutes
  Simple mask at 60 L/min: After 3 minutes of oxygen supplementation (preoxygenation), with each of the devices listed in the arms above, the exhaled oxygen content will be measured.
- Non-rebreather at 15 L/Min: Non-rebreather at 60 L/min
  Non-rebreather at 15 L/min: After 3 minutes of oxygen supplementation (preoxygenation), with each of the devices listed in the arms above, the exhaled oxygen content will be measured.
- Non-rebreather at 60 L/Min: Non-rebreather at 60 L/min for 3 minutes
  Non-rebreather at 60 L/min: After 3 minutes of oxygen supplementation (preoxygenation), with each of the devices listed in the arms above, the exhaled oxygen content will be measured.
- Bag Valve Mask at 15 L/Min: Bag valve mask at 15 L/min for 3 minutes
  Bag valve mask at 15 L/min: After 3 minutes of oxygen supplementation (preoxygenation), with each of the devices listed in the arms above, the exhaled oxygen content will be measured.
Arm/Group | Simple Mask | Non-rebreather at 15 L/Min | Non-rebreather at 60 L/Min | Bag Valve Mask at 15 L/Min
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No